CLINICAL TRIAL: NCT03750539
Title: Phase II Randomized Study of Concurrent Chemotherapy and Pelvic Radiation Therapy With Standard Fractionated Compared to Hypofractionated Followed by Surgery for Patients With Locally Advanced Cervical Cancer.
Brief Title: Chemotherapy and Pelvic Hypofractionated Radiation Followed by Surgery Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Principal Investigator, David Cantu, Chief of clinical trial departament, National Institute of Cancerología
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 017/020/ICI
Record Dates: First submitted 2018-11-05; First posted 2018-11-23 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiation Dose Hypofractionation; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Phase II Comparative Randomized Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment (Active Comparator): External Beam pelvic radiation therapy daily dose of 1.8-2 Gray (Gy) per session for 25 sessions to accomplish 45 Gy Chemotherapy ( cisplatin 40mg/m2), intravenous administration of chemotherapy once a week in an hour infusion Type II or type III open radical hysterectomy after 4-6 weeks after completion of external beam radiation
  Interventions: Radiation: Standard radiotherapy; Procedure: Radical hysterectomy
- hypofractionated treatment (Experimental): External Beam pelvic radiation therapy daily dose of 1.8-2gy per session for 15 sessions to accomplish 37.5 Gy Chemotherapy ( cisplatin 40mg/m2), intravenous administration of chemotherapy once a week in an hour infusion Type II or type III open radical hysterectomy after 4-6 weeks after completion of external beam radiation
  Interventions: Radiation: hypofractionated radiotherapy; Procedure: Radical hysterectomy

INTERVENTIONS:
Radiation: Standard radiotherapy — External Bean Pelvic Radiation: 50 Gy in 15 fractions, with weekly cisplatin.
  Arms: Standard Treatment
Radiation: hypofractionated radiotherapy — External Bean Pelvic Radiation: 37.5 Gy in 15 fractions, with weekly cisplatin.
  Arms: hypofractionated treatment
Procedure: Radical hysterectomy — Radical hysterectomy and pelvic and paraaortic lymph node resection
  Other Names: Surgery

SUMMARY:
The purpose of the study is to evaluate the role of hypofractionated in the treatment of locally advanced cervical cancer. The study will be conducted in Honduras and Mexico, and patients will be randomized to a standard fraction (45 Gy in 25 fractions) or hypofractionated (37.5Gy in 15 fractions) followed by surgery. Patients will receive weekly cisplatin with their treatments at 40 mg/m2. Response rate, survival, and toxicity will be evaluated.

DETAILED DESCRIPTION:
Toxicity will be assessed six times during this study. In addition to the primary endpoint of patient-reported gastrointestinal toxicity, a broad range of other toxicities will be comprehensively evaluated, including urinary, hematologic and dermatologic, this data will allow to determining the effect of hypofractionated radiation therapy on each of these aspects of toxicity from pelvic radiation. Additionally, will be recognized that it is possible to advance in the understanding of the clinical risk and benefits of hypofractionation.

The primary endpoint will be acute gastrointestinal toxicity using the Radiation Therapy Oncology Group (RTOG) common toxicity criteria.

In total, evaluating toxicity in different time points will allow determining if hypofractionation is secure concerning acute and late toxicity, that would enable to offer an optional treatment to this kind of patient. Chronic gastrointestinal toxicity from radiation continues to increase rapidly over two years, and then the rate of developing new toxicities slows. As a result, the majority of chronic radiation-induced gastrointestinal toxicity by evaluating toxicity two years after completion of radiotherapy is going to be identified.

Quality of life (QOL) will be evaluated using EORTC QLQ-CX24 and EORTC QLQ-C30, both of which have been validated and available in Mexican Spanish.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have International Federation of Gynecology and Obstetrics (FIGO) stage IB2-IIB squamous, adenosquamous or adenocarcinoma of cervical with no disease outside of the pelvis by via ultrasound.
* No distant metastasis via chest X-ray.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Age 18
* complete blood count (CBC)/differential obtained 14 days before study entry with adequate bone marrow function defined as follows:
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mim3
* Platelets 100,000 cells/mim3
* Hemoglobin 8.0 g/dl
* White blood count 4000 cell/m3
* An adequate renal function defined as follows:
* Serum creatinine 1.5 mg/dl within 14 days before study entry
* Patients with known HIV positive must have a cluster of differentiation 4 (CD4) T lymphocytes count be 350 cells/mm3 within 14 days prior to study entry (note, however, that HIV testing is not required for entry into this protocol). Excluding HIV positive patients with invasive cervical cancer and low CD4 cell counts is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
* Chest x-ray and ultrasound must be performed within 12 (8 or 12) weeks before the study enrollment (I took out the ct scan of abdomen and pelvis)
* Patient must provide study-specific informed consent before study entry.

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (For example, carcinoma in situ of the breast or oral cavity.
* Patients cannot have any neuroendocrine histology in pathology.
* Prior systemic chemotherapy for the current cervical cancer, note that prior chemotherapy for a different cancer is allowable.
* Prior radiation therapy to the pelvis that would result in overlap of radiation therapy fields.
* Severe active co-morbidity, defined as follows:
* Unstable angina or congestive heart failure requiring hospitalization within the last six months.
* Transmural myocardial infarction within the previous six months.
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of the study entry.
* Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of study entry.
* Coagulation defects; note, however, that coagulation parameter are not required for entry into this protocol.
* Prior allergic reaction to cisplatin or other platinum drugs.
* Patients with para-aortic nodes or distant metastasis.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-10 (Actual); Primary Completion 2024-11-10 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Acute and late toxicity. | 2 years
  Number of Participants With Treatment-Related Adverse Events as Assessed by RTOG

SECONDARY OUTCOMES:
Overall survival | 2 years
  Number of Participants dead at two years according to kaplan-meyer analysis
disease specific survival | 2 years
  Number of Participants dead of disease at two years according to kaplan-meyer analysis
equivalent treatment | 2 years
  hypofractionated radiotherapy is similar in toxicity and disease control compared to standard external beam treatment.
Surgical complications | 1 year
  comparison of surgical complications between the two arms of treatment according to The Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: David F Cantu-de Leon, MD, Msc, PhD, Principal Investigator — Instituto Nacional de Cancerologia, Columbia
Locations (2):
- Mexico (2):
  - David Cantu de Leon, Mexico City, Tlalpan
  - Instituto Nacional de Cancerologia, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: the data will be shared with scientific and academic institutions or research groups that study the same topic and with the regulatory and ethical authorities that require it, to ensure the quality and accuracy of the data.